CLINICAL TRIAL: NCT00424788
Title: A Multicenter Study to Assess the Effect of Plasma Exchange in Accelerating the Clearance of Natalizumab in Subjects With Multiple Sclerosis (MS)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101MS001
Record Dates: First submitted 2007-01-18; First posted 2007-01-22 (Estimated); Last update posted 2009-09-04 (Estimated); Status verified 2009-09

CONDITIONS: Relapsing Forms of Multiple Sclerosis
Keywords: multiple sclerosis (MS)
MeSH Terms: conditions — Multiple Sclerosis | interventions — Plasma Exchange

INTERVENTIONS:
Procedure: Plasma exchange
Drug: natalizumab treatment

SUMMARY:
Natalizumab (TYSABRI) is a protein-based drug that is manufactured by Biogen Idec in partnership with Elan Pharmaceuticals. Natalizumab is approved in the US and Europe for the treatment of Multiple Sclerosis (MS). The purpose of this study is to determine whether the amount of natalizumab (TYSABRI) that is present in your blood (plasma) can be reduced or eliminated by separating and removing the plasma and replacing it with other fluids, a process called plasma exchange.

ELIGIBILITY:
Inclusion Criteria:

* considered by the Investigator to be free of signs and symptoms suggestive of any serious opportunistic infection
* willing to discontinue and remain free from concomitant immunosuppressive or immunomodulatory treatment (including interferon beta and glatiramer acetate) for the duration of the study
* willing and able to comply with the site's plasma exchange protocol which may require hospitalization or daily visits

Exclusion Criteria:

* considered by the Investigator to be immunocompromised
* history of, or available abnormal laboratory results indicative of any major disease that would preclude the administration of a recombinant humanized antibody immunomodulating agent for the duration of the study.
* condition(s) considered to be contraindication(s) for plasma exchange, including but not limited to bleeding diathesis, hypotension, or vascular access limitations

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2007-01; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Panzara, MD MPH, Study Director — Biogen
Locations (2):
- United States (2):
  - Cleveland Clinic Mellen Center for MS, Cleveland, Ohio
  - Center for Neurological Disorders, Aurora Health Care, Milwaukee, Wisconsin